CLINICAL TRIAL: NCT00874315
Title: A Multicenter Pilot Study of Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation With In-vivo T-cell Depletion to Evaluate the Role of NK Cells and KIR Mis-matches in Relapsed or Refractory High-risk Neuroblastoma.
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation for Relapsed or Refractory High-Risk NBL.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000636111; NCH-08-0234 (Registry Identifier: Nationwide Children's Hospital IRB); IRB-2008-0230 (Registry Identifier: National Marrow Donor Program IRB)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Neuroblastoma
Keywords: recurrent or refractory neuroblastoma
MeSH Terms: conditions — Neuroblastoma; Recurrence | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: anti-thymocyte globulin — 2.5 mg/kg/day for 4 doses on day -3, -2 , -1 and day +2.
  Other Names: Thymoglobulin
Drug: busulfan — 0.8 mg/kg/dose for total of 8 doses.
  Other Names: Busulfex
Drug: cyclosporine — 1.5 mg/kg/dose every 12 hours.
  Other Names: Sandimmune, Gengraf, Neoral.
Drug: fludarabine phosphate — 30 mg/m2/day for 5 days.
  Other Names: Fludara
Drug: mycophenolate mofetil — 15 mg/kg/dose every 8 hours
  Other Names: Cell-cept
Drug: tacrolimus — 0.03 mg/kg/day as continuous infusion or 12 hour divided doses
Procedure: allogeneic hematopoietic stem cell transplantation — Donor stem cell transplantation from HLA matched sibling donor or an unrelated donor.

SUMMARY:
RATIONALE: - Relapsed or refractory Neuroblastoma (NBL) carries a very poor prognosis and children with relapsed NBL have an overall 3 year survival rate of < 10%. Hematopoietic Stem Cell Transplant from a different donor (allogeneic), is a form of adoptive cellular therapy , such that infused donor cells find host tumors as foreign and fight them. After transplant, the donor immune cells (i.e. T cells, NK cells) mediate Graft versus Tumor (GVT) effect and may stop tumor from recurring. Also,reduced intensity transplants lead to minimal toxicity and less risk of mortality in heavily pre-treated NBL patients.

PURPOSE: This phase II trial is studying how well giving a reduced intensity(using Fludarabine, Busulfan and antithymocyte globulin)preparative regimen followed by donor stem cell transplant works in treating young patients with high-risk neuroblastoma that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility of allogeneic hematopoietic stem cell transplantation after a reduced-intensity conditioning regimen comprising fludarabine phosphate, busulfan, and anti-thymocyte globulin, in terms of donor engraftment, transplant-related mortality, and development of acute and chronic graft-vs-host disease, in pediatric patients with high-risk relapsed or refractory neuroblastoma.

Secondary

* To elucidate the role of natural killer (NK) cells as effectors of graft-vs-tumor effect in these patients.
* To evaluate the role of killer immunoglobulin-like receptor (KIR) mismatches in the donor-recipient pairs on the outcomes of these patients.
* To determine the incidence of progression-free survival at 1 year post-transplantation in these patients.

OUTLINE: This is a multicenter study.

* Reduced-intensity conditioning regimen: Patients receive fludarabine phosphate IV over 1 hour on days -10 to -6, busulfan IV over 2 hours once on day -10 (test dose) and then every 6 hours on days -5 and -4, and anti-thymocyte globulin IV over 6-8 hours on days -3 to -1 and on day 2.
* Transplantation: Patients undergo allogeneic bone marrow or G-CSF-mobilized peripheral blood stem cell transplantation on day 0.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive cyclosporine or tacrolimus IV or orally beginning on day -2 and continuing until day 60 or day 100, followed by a taper until day 100 or day 180 in the absence of GVHD. Patients also receive mycophenolate mofetil IV or orally on days 1-30, followed by a taper until day 60 in the absence of GVHD.

Blood samples are collected at baseline and on days 30, 60, and 100 for correlative laboratory studies. Samples are analyzed for killer immunoglobulin-like receptor (KIR) mismatches by genotyping and immunophenotyping methods (PCR and flow cytometry); natural killer (NK) cell reconstitution by flow cytometry; and NK cell function, NK cell allo-reactivity by ELISPOT and ELISA.

After completion of study treatment, patients are followed periodically for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of high-risk neuroblastoma, meeting one of the following criteria:

  * Refractory disease, defined as no response, mixed response, or progressive disease after completion of induction therapy administered according to clinical trials COG-A3973 or COG-ANBL0532 (or other similar high-intensity induction regimen)
  * Relapsed following high-dose chemoradiotherapy including autologous stem cell transplantation
* Achieved a complete remission (CR), very good partial remission (VGPR), or partial remission (PR) after ≤ 2 different salvage regimens, as defined by the following:

  * In CR after treatment with some form of salvage therapy (e.g., ¹³¹I-MIBG, antibody-based therapy, or any other COG or NANT salvage-therapy regimen)
  * In VGPR or PR after salvage therapy

    * No more than 3 sites of skeletal disease as determined by an ¹²³I-MIBG scan (for regional involvement of the skeleton [e.g., pelvis, spine], the tumor involvement should be < 25% of the site)
    * Bone marrow involvement (< 25% neuroblasts) by morphologic exam within the past 2 weeks
    * Patients with soft tissue disease are eligible provided they exhibit either a VGPR or PR in the primary soft tissue mass and in any sites of metastatic soft tissue disease
* Disease status meeting one of the following criteria:

  * Minimal residual disease
  * Disease considered responsive to a salvage regimen
  * Stable disease
* No rapidly progressive disease
* Donors must meet one of the following criteria:

  * Matched, related donor (6/6 or 5/6) (bone marrow donor allowed)
  * HLA-matched unrelated donor (10/10 match on high-resolution [HR] typing of HLA-A, B, C, DRB1, and DQB1)
  * One allele- or antigen-mismatched unrelated donor (9/10 match on HR typing), mismatched at HLA-C only
  * One allele- or antigen-mismatched unrelated donor (9/10 match on HR typing), mismatched at HLA-A, B, DRB1, or DQB1 (only when HLA-C mismatch is not available)

PATIENT CHARACTERISTICS:

* Karnofsky/Lansky performance status 60-100%
* ANC > 500/mm^3
* Creatinine clearance or radioisotope GFR ≥ 60 mL/min
* Total bilirubin < 3.0 mg/dL
* AST or ALT < 5 times upper limit of normal
* Shortening fraction ≥ 25% by ECHO OR ejection fraction > 30% by MUGA
* FEV_1 and DLCO ≥ 30% OR normal chest x-ray, pulse oximetry, and venous blood gas
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active or recent (within the past 30 days) fungal infection
* No proven or suspected sepsis, pneumonia, or meningitis unless appropriate therapeutic measures have been initiated to control the infection and systemic signs are no longer life-threatening
* No requirement for oxygen or ventilator support

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior tandem autologous stem cell transplantations (according to clinical trial COG-ANBL0532) allowed
* No prior allogeneic hematopoietic stem cell transplantation
* More than 2 months since prior autologous stem cell transplantation, myeloablative therapy, total-body irradiation, whole abdominal radiotherapy, or therapeutic ¹³¹I-MIBG
* More than 3 weeks since prior chemotherapy, immunotherapy (including anti-GD2 regimen), or biologic response modifiers and recovered
* More than 2 weeks since prior local radiotherapy to the sites of metastatic disease

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by the incidence of donor engraftment, transplant-related mortality, and grade III-IV acute graft-vs-host disease (GVHD) at day 100 and the incidence of extensive chronic GVHD within the first year post-transplantation | 100 days post-HSCT
  The safety and feasibility of reduced intensity allogeneic HSCT will be established in this population by monitoring the incidence of adverse events- 100 day mortality,incidence of severe acute GVHD and non-engraftment of donor cells.

SECONDARY OUTCOMES:
Progression-free survival (PFS) at 1 year | 1 year post- HSCT
Relationship between biologic endpoints (e.g., number of natural killer [NK] cells infused, NK cell recovery, and NK cell chimerism status) and clinical endpoints (e.g., donor engraftment, acute GVHD, transplant-related mortality, and PFS) | 3 and 6 months post-SCT
Relationship between presence of killer immunoglobulin-like receptor (KIR) mismatches and clinical endpoints | 3 and 6 months post-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Soni, MD, Principal Investigator — Nationwide Children's Hospital
Locations (4):
- United States (4):
  - Children's Memorial Hospital, Chicago, Illinois
  - Morgan Stanley Children's Hospital of NY, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hopsital of Wisconsin, Milwaukee, Wisconsin